CLINICAL TRIAL: NCT06332599
Title: Minocycline-containing Bismuth Quadruple Therapy for Helicobacter Pylori Rescue Treatment: a Real-world Evidence Study
Brief Title: Minocycline for Helicobacter Pylori Rescue Treatment
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, RenJi Hospital
Other Study IDs: rjhy20240001
Record Dates: First submitted 2024-03-17; First posted 2024-03-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; rescue therapy; minocycline
MeSH Terms: conditions — cyclopia sequence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- BQT
  Interventions: Drug: BQT
- PBM4M4
  Interventions: Drug: PBM4M4
- PBM3M3
  Interventions: Drug: PBM3M3
- PBM2M4
  Interventions: Drug: PBM2M4
- PBM2M3
  Interventions: Drug: PBM2M3

INTERVENTIONS:
Drug: BQT — PPI（esomeprazole or vonoprazan) 20 mg twice daily, bismuth potassium citrate 600 mg (220 mg elemental bismuth) twice daily, tetracycline 500 mg four times a day, and metronidazole 400 mg four times a day
  Groups: BQT
Drug: PBM4M4 — PPI（esomeprazole or vonoprazan) 20 mg twice daily, bismuth potassium citrate 600 mg (220 mg elemental bismuth) twice daily, minocycline 50 mg four times a day, and metronidazole 400 mg four times a day
  Groups: PBM4M4
Drug: PBM3M3 — PPI（esomeprazole or vonoprazan) 20 mg twice daily, bismuth potassium citrate 600 mg (220 mg elemental bismuth) twice daily, minocycline 50 mg three times a day, and metronidazole 400 mg three times a day
  Groups: PBM3M3
Drug: PBM2M4 — PPI（esomeprazole or vonoprazan) 20 mg twice daily, bismuth potassium citrate 600 mg (220 mg elemental bismuth) twice daily, minocycline 50 mg twice daily, and metronidazole 400 mg four times a day
  Groups: PBM2M4
Drug: PBM2M3 — PPI（esomeprazole or vonoprazan), bismuth potassium citrate 600 mg (220 mg elemental bismuth) twice daily, minocycline 50 mg twice daily, and metronidazole 400 mg three times a day
  Groups: PBM2M3

SUMMARY:
Current guidelines have recommended classical bismuth-containing quadruple therapy including proton-pump inhibitor, bismuth, tetracycline, metronidazole as the empirical rescue therapy. However, tetracycline is clinically unavailable in China and the high frequency of adverse events of bismuth quadruple therapy often result in poor compliance, which limited the applicability of this recommendation. We previously showed that the efficacy of bismuth-containing quadruple therapy with minocycline and metronidazole was not inferior to classical bismuth quadruple therapy for refractory H. pylori infection, though also accompanied with high occurrence of adverse events.This study aimed to evaluate the efficacy and tolerability of four different regimens with minocycline and metronidazole compared to classical bismuth quadruple therapy for H. pylori rescue treatment in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed H. pylori infection and with previous treatment failure

Exclusion Criteria:

* subjects naive to H. pylori treatment,
* history of gastrectomy
* pregnant or lactating women
* severe systemic diseases or malignancy
* administration of antibiotics, bismuth, antisecretory drugs, or Chinese herb medicine in the preceding 12 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who failed at least two courses of H. pylori treatment containing clarithromycin, nitroimidazoles, fluoroquinolones, and/or amoxicillin, and received 14-day tetracycline/minocycline, metronidazole-containing bismuth quadruple therapy were identified. Patients with the following criteria were excluded: (1) naive to H. pylori treatment; (2) under 18 or over 80 years; (3) history of gastrectomy; (4) administration of antibiotics, bismuth, acid suppressants, or Chinese herb medicine in the preceding 12 weeks; (5) severe systemic diseases or malignancy.
Sampling Method: Probability Sample
Enrollment: 823 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within six weeks after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities)
Compliance rate | Within six weeks after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, None Selected, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Y, Qiu S, Guo Y, Chen J, Li M, Ding Z, Zhang W, Liang X, Lu H. Optimization of Minocycline-Containing Bismuth Quadruple Therapy for Helicobacter pylori Rescue Treatment: A Real-World Evidence Study. Helicobacter. 2024 Sep-Oct;29(5):e13138. doi: 10.1111/hel.13138. PMID 39306798